CLINICAL TRIAL: NCT04915690
Title: Investigation on the Practice Status of Emergency Doctors and Nurses
Brief Title: Investigation on the Practice Status of Emergency Stuff
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Hospital (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Litongde Hospital (Unknown); Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Children's Hospital Affiliated to Zhejiang University School of Medicine (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Traditional Chinese Medicine Hospital (Unknown); The Third Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine (Unknown); The 90th and Third Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army (Unknown); The 72nd Group Army Hospital of the Chinese People's Liberation Army (Unknown); Zhejiang Provincial Hospital of the Chinese People's Armed Police Force (Unknown); First People's Hospital of Hangzhou (Other); The Third People's Hospital of Hangzhou (Other); Red Cross Hospital, Hangzhou, China (Other); Hangzhou Traditional Chinese Medicine Hospital (Unknown); The Affiliated Hospital of Hangzhou Normal University (Other); Hangzhou Dajiangdong Hospital (Unknown); The First People's Hospital of Xiaoshan District (Unknown); Hangzhou Xiaoshan Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Yuhang District (Other); The Second People's Hospital of Yuhang District (Unknown); The Third People's Hospital of Yuhang District (Unknown); Yuhang Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Fuyang District (Unknown); Fuyang District Traditional Chinese Medicine Hospital (Unknown); Lin'an People's Hospital (Unknown); Lin'an Traditional Chinese Medicine Hospital (Unknown); The First People's Hospital of Tonglu County (Unknown); Tonglu Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Chun'an County (Unknown); Chun'an County Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Jiande City (Unknown); Jiande City Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Huzhou (Other); Huizhou Municipal Central Hospital (Other); Huzhou Traditional Chinese Medicine Hospital (Unknown); Huzhou Third People's Hospital (Other); People's Hospital of Wuxing District, Huzhou City (Unknown); People's Hospital of Nanxun District, Huzhou City (Unknown); Anji County People's Hospital (Unknown); The Third People's Hospital of Anji County (Unknown); Deqing County People's Hospital (Unknown); Changxing People's Hospital (Other); Changxing County Hospital of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jiaxing Traditional Chinese Medicine Hospital (Unknown); Haining People's Hospital (Unknown); Haining Traditional Chinese Medicine Hospital (Unknown); The First People's Hospital of Tongxiang City (Unknown); Haiyan County People's Hospital (Unknown); The First People's Hospital of Jiashan County (Unknown); Jiashan County Hospital of Traditional Chinese Medicine (Unknown); Zhejiang Xin'an International Hospital (Unknown); Jinhua Central Hospital (Other); Jinhua City People's Hospital (Unknown); Jinhua Traditional Chinese Medicine Hospital (Unknown); The First People's Hospital of Wucheng District, Jinhua City (Unknown); People's Hospital of Wucheng District, Jinhua City (Unknown); Second People's Hospital of Jindong District, Jinhua City (Unknown); Yiwu Central Hospital (Other); Dongyang People's Hospital (Other); Dongyang Traditional Chinese Medicine Hospital (Unknown); Lanxi People's Hospital (Other); Lanxi Traditional Chinese Medicine Hospital (Unknown); Hangzhou Medical College (Other); Yongkang Traditional Chinese Medicine Hospital (Unknown); Pujiang County People's Hospital (Unknown); Pujiang County Hospital of Traditional Chinese Medicine (Unknown); Pan'an County People's Hospital (Unknown); The First People's Hospital of Wuyi County (Unknown); The Sixth Affiliated Hospital of Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); Lishui Traditional Chinese Medicine Hospital (Unknown); Liandu District People's Hospital (Unknown); Longquan People's Hospital (Unknown); Jinyun County People's Hospital (Unknown); Jingning County People's Hospital (Unknown); Qingtian County People's Hospital (Unknown); Qingyuan People's Hospital (Other); Songyang County People's Hospital (Unknown); Songyang County Hospital of Traditional Chinese Medicine (Unknown); Suichang County People's Hospital (Unknown); Yunhe County People's Hospital (Unknown); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); Ningbo Third Hospital (Unknown); Li Huili Hospital, Ningbo Medical Center (Unknown); Ningbo Traditional Chinese Medicine Hospital (Unknown); Ningbo Ninth Hospital (Unknown); People's Hospital of Beilun District, Ningbo City (Unknown); Ningbo Yinzhou People's Hospital (Unknown); The Second Hospital of Yinzhou District, Ningbo City (Unknown); The Second Hospital of Haishu District, Ningbo City (Unknown); People's Hospital of Zhenhai District, Ningbo City (Unknown); People's Hospital of Fenghua District, Ningbo City (Unknown); Ningbo Women & Children's Hospital (Other); Mingzhou Hospital of Zhejiang University (Unknown); Yuyao People's Hospital (Other); Cixi City People's Hospital (Unknown); Ninghai County First Hospital (Unknown); Xiangshan County First People's Hospital Medical and Health Group (Unknown); People's Hospital of Quzhou (Other); Quzhou Second People's Hospital (Unknown); Zhejiang Quhua Hospital (Other); Quzhou Traditional Chinese Medicine Hospital (Unknown); People's Hospital of Kecheng District, Quzhou City (Unknown); Jiangshan City People's Hospital (Unknown); Jiangshan Traditional Chinese Medicine Hospital (Unknown); Jiangshan Beilin Hospital (Unknown); Kaihua County People's Hospital (Unknown); Kaihua County Hospital of Traditional Chinese Medicine (Unknown); Changshan County People's Hospital (Unknown); Longyou County People's Hospital (Unknown); Longyou County Hospital of Traditional Chinese Medicine (Unknown); Shaoxing People's Hospital (Other); Shaoxing Central Hospital (Other); Shaoxing Second Hospital (Other); Shaoxing Traditional Chinese Medicine Hospital (Unknown); Shangyu People's Hospital of Shaoxing City (Unknown); Shangyu Hospital of Traditional Chinese Medicine, Shaoxing City (Unknown); Traditional Chinese Medicine Hospital of Keqiao District, Shaoxing City (Unknown); Zhuji City People's Hospital (Unknown); Zhuji City Hospital of Traditional Chinese Medicine (Unknown); Shengzhou Traditional Chinese Medicine Hospital (Unknown); Xinchang County People's Hospital (Unknown); Taizhou Hospital (Other); Taizhou Enze Medical Center Group (Other); Taizhou First People's Hospital (Other); Taizhou Hospital of Traditional Chinese Medicine (Other Government); Second People's Hospital of Linhai City (Unknown); First People's Hospital of Linhai City (Unknown); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Wenling Traditional Chinese Medicine Hospital (Unknown); Yuhuan City People's Hospital (Unknown); Sanmen County People's Hospital (Unknown); Tiantai County People's Hospital (Unknown); Xianju County People's Hospital (Unknown); Wenzhou Central Hospital (Other); Wenzhou People's Hospital (Other); Wenzhou Traditional Chinese Medicine Hospital (Unknown); Wenzhou Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Lucheng District People's Hospital of Wenzhou City (Unknown); The First People's Hospital of Longwan District, Wenzhou City (Unknown); Wenzhou Longwan District Integrated Traditional Chinese and Western Medicine Hospital (Unknown); Wenzhou Ouhai District People's Hospital (Unknown); The Third People's Hospital of Ouhai District, Wenzhou City (Unknown); Wenzhou Ouhai District Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Wenzhou Dongtou District People's Hospital (Unknown); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); The Second People's Hospital of Yueqing City (Unknown); The Third People's Hospital of Yueqing City (Unknown); The Fifth People's Hospital of Yueqing City (Unknown); Yueqing Traditional Chinese Medicine Hospital (Unknown); The Third Affiliated Hospital of Wenzhou Medical University (Other); Ruian City Hospital of Traditional Chinese Medicine (Unknown); Longgang People's Hospital (Unknown); Cangnan County People's Hospital (Unknown); The Third People's Hospital of Cangnan County (Unknown); Cangnan County Hospital of Traditional Chinese Medicine (Unknown); Pingyang County People's Hospital (Unknown); Second People's Hospital of Pingyang County (Unknown); Pingyang County Hospital of Traditional Chinese Medicine (Unknown); Taishun County People's Hospital (Unknown); Taishun County Hospital of Traditional Chinese Medicine (Unknown); Yongjia County People's Medical Hospital (Unknown); Yongjia County Hospital of Traditional Chinese Medicine (Unknown); Wencheng County People's Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Zhoushan Traditional Chinese Medicine Hospital (Unknown); Zhoushan Women and Children's Hospital (Unknown); Central Hospital of Dinghai District, Zhoushan City (Unknown); Putuo Hospital (Unknown); The First People's Hospital of Daishan County (Unknown); Shengsi County People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-0292
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Emergencies
Keywords: Emergency department; practice status; doctors and nurses
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is the medical environment of the emergency department? Is the practice status of emergency medical care good or bad? At present, there is no corresponding investigation and research on the current situation of emergency medical care in China. Therefore, this study intends to conduct a cross-sectional survey of the current practice of emergency medical staff to understand the current situation of emergency medical care and provide a basis for the development and construction of the emergency department.

DETAILED DESCRIPTION:
As the window department of the hospital, the emergency department is an important place for the rescue of critically ill patients. Whether the emergency department can complete the rescue of various critically ill patients with high standards, high efficiency and high quality reflects the overall management level and technical capabilities of the hospital. With the development of society, the people's demand for emergency medical services is also increasing. Therefore, it is important to strengthen the investment of manpower and material resources in the emergency department. Since the outbreak of the new crown pneumonia epidemic, the emergency department has been the frontier of contact with the epidemic, and the busy emergency patients have faced greater risks and challenges. So, what is the medical environment of the emergency department? Is the practice status of emergency medical care good or bad? At present, there is no corresponding investigation and research on the current situation of emergency medical care in China. Therefore, this study intends to conduct a cross-sectional survey of the current practice of emergency medical staff to understand the current situation of emergency medical care and provide a basis for the development and construction of the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All hospitals with independent emergency departments in Zhejiang Province;
* Voluntary participation.

Exclusion Criteria:

* hospitals without independent emergency department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Doctors and nurses who work within the scope of the survey and meet the criteria for inclusion in the emergency department of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
General information and working conditions survey | 1 month
  Gender, age, hospital grade, job title, working hours, work department
Working hours and income survey | 1 month
  Weekly working hours, night shift frequency, rest time, annual rest time, income situation, income satisfaction
Practice environment and medical violence survey | 1 month
  Practice environment, medical violence experience
Continuing education and career prospects survey | 1 month
  Continuing education, learning opportunities, promotion of professional titles, promotion pressure, career prospects
Health status and work attitude survey | 1 month
  Health status, disease status, attitude towards work

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, MD, Study Chair — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China